CLINICAL TRIAL: NCT05956197
Title: Efficacy of High Dose Albumin Therapy in Improving Liver Transplant-free Survival in Patients With Acute Decompensation of Cirrhosis- A Prospective Cohort Study
Brief Title: Efficacy of High Dose Albumin Therapy in Improving Liver Transplant-free Survival in Patients With Acute Decompensation of Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-50
Record Dates: First submitted 2022-06-18; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Decompensation of Cirrhosis: Acute Decompensation of Cirrhosis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. This is a cohort study

SUMMARY:
Research Objectives- We hypothesized high-dose 25% albumin would be superior to standard medical treatment in improving 3-month mortality in patients with acute decompensation of cirrhosis by improving the systemic hemodynamics and amelioration of systemic inflammation, endothelial function and coagulation.

Aim: To study the efficacy of 25% albumin in reducing 3-month mortality in acute decompensation in cirrhosis.

Primary Objective

• To study the efficacy of 25% albumin in reducing the 3-month mortality.

Secondary Objectives

* To study the cumulative incidence of liver related complications (paracentesis induced circulatory dysfunction (PICD), AKI, hyponatremia, hepatic encephalopathy and variceal bleed)
* Improvement in MELD, CTP, SOFA and AARC scores
* Impact on cardiac function and systemic hemodynamics
* Impact of albumin on development of SBP and non-SBP infections
* Survival free of liver transplant and TIPS at 3 months
* Effect of albumin therapy on immunomodulation, dysfunctional albumin, endothelial function and coagulation at 3 months
* Proportion of patients achieving recompensation at 3 months
* Time to achieve serum albumin >4 g/dL and its correlation with clinical outcomes.

DETAILED DESCRIPTION:
Methodology

DOSING REGIMEN In this prospective cohort study, consecutive cirrhotic patients, fulfilling the inclusion criteria and exclusion criteria will be enrolled. Details of sample size calculation are given under section of statistical methods. Severity of liver disease will be assessed according to severity scores- CTP and MELD score.

The patients will be enrolled and administered high dose 25% albumin at 1.5 gm/kg/week for 12 weeks and subsequently followed for development of liver related complications, need of hospitalizations and paracentesis. The impact of albumin therapy on systemic hemodynamics, cardiac function, systemic inflammation, bacterial infections and endothelial function and coagulation will be studied. Patients would be given standard medical treatment as per the institutional protocol.

Important definitions:

Acute decompensation of cirrhosis will be defined according to the APASL criteria. This occurs in a cirrhotic with or without prior decompensation and is often associated with a precipitant. The presentation of AD is either hepatic (jaundice, ascites, HE) or extrahepatic (variceal bleed, acute kidney injury or sepsis), and time period is up to 3 months.

Infections: would be defined as under Pneumonia: Newly acquired respiratory symptoms (cough, sputum production and/or dyspnea) and chest radiography showing lung infiltrate [2] Spontaneous bacteremia: Positive blood cultures with no cause of bacteremia [2] Urinary tract infection: More than 10 leukocytes per high-power field in urine and positive urine cultures [3] Spontaneous Bacterial Peritonitis: Was diagnosed in the presence of ascitic fluid neutrophil count >250mm3 [7] Hepatic encephalopathy: Was defined as per the West-Haven's criteria [5] Acute variceal bleed: Was diagnosed as per Baveno V endoscopic criteria [6] Refractory/Recurrent ascites: As per the EASL criteria [8] Paracentesis Induced Circulatory Dysfunction: PICD was defined as a 50% increase in PRA over baseline on day 6. [9] Acute Kidney Injury: Would be defined according to the IAC criteria [10] Recompensation: defined as decompensated patients (previous episode of ascites) that were clinically inapparent without ascites or with controlled ascites using medical treatment at time of inclusion. [11]

Investigations: Baseline HVPG with assessment of portal (systemic and pulmonary hemodynamics) and cardiac reserve systolic and diastolic function (2D-ECHO and stress echocardiography), cystatin C, urine NGAL and KIM-1, plain CT, cardiac biomarkers (NT-Pro BNP, Troponin I), albumin isoforms, cytokine array, endotoxin levels. Markers of endothelial function (ADAMTS, vWF) and coagulation (rotational thromboelastometry EXTEM) Plain CT-scan for assessment of sarcopenia, body composition analysis. Body weight, blood pressure and stress echocardiogram (if feasible) would be done for all patients. Glomerular filtration rate (GFR) will be estimated by using eGFR equations -modification of diet in renal disease (MDRD6) and Cystatin C based (Chronic kidney disease Epidemiology Collaboration). Along with this, arterial blood sample will be collected after overnight fast and bed rest at least for 8 h in supine position for plasma renin activity, plasma aldosterone and plasma norepinephrine concentration. Patients would subsequently undergo HVPG, cystatin C, cardiac function, cardiac biomarkers (NT-Pro BNP and Troponin I), cytokine profile, albumin isoforms at 3 months and 6 months. A repeat plain CT scan to assess sarcopenia would be done at 3 months and at 6 months. The follow up would be 1 year or until TIPS or liver transplant.

Assessment of cardiac function: This can be assessed as systolic or diastolic dysfunction.Systolic dysfunction will be defined as a blunted increase in cardiac output on exercise, volume challenge or pharmacological stimuli or resting ejection fraction <55 %.

Diastolic dysfunction will be defined according to the ratio of early to late (atrial) phases of ventricular filling or E/A ratio <1.0 (age-corrected), prolonged deceleration time (>200 ms), or prolonged isovolumetric relaxation time (>80 ms) Dobutamine stress echocardiography(DSE)-The left ventricular(LV) systolic and diastolic functions will be evaluated by two-dimensional and Doppler echocardiography at rest and during peak dobutamine infusion (40 µg/kg/min). An abnormal response will be defined as a decrease of less than 10% in LV end-diastolic volume, a decrease of less than 20% in end-systolic volume, and an increase of less than 10% in LV ejection fraction (EF) at peak dobutamine infusion Chronotropic incompetence-Heart rate reserve (HRR) will be measured by the formula (HRR)={[(peak HR-HR at rest)/(220-age-HR at rest)]×100} .Chronotropic incompetence will be defined as HRR less than 80%.

Diastolic dysfunction occurs when the left ventricular myocardium is non-compliant and not able to accept blood return in a normal fashion from the left atrium. There are four grades of diastolic dysfunction as described below. Echocardiography is the gold standard to diagnose diastolic dysfunction.

Grade I Diastolic dysfunction :This is a normal finding and occurs in nearly 100% of individuals by the age of 60. The E wave velocity is reduced resulting in E/A reversal (ratio < 1.0). The left atrial pressures are normal. The deceleration time of the E wave is prolonged measuring > 200 ms. The e/e' ratio measured by tissue Doppler is normal.

Grade II diastolic dysfunction:This is pathological and results in elevated left atrial pressures. The E/A ratio is normal (0.8 +- 1.5), the deceleration time is normal (160-200 ms), however the e/e' ratio is elevated. The E/A ratio will be < 1 with Valsalva. A major clue to the presence of grade II diastolic dysfunction as compared to normal diastolic function is the presence of structural heart disease such as left atrial enlargement, left ventricular hypertrophy or systolic dysfunction.

Grade III Diastolic dysfunction :This results in significantly elevated left atrial pressures. Also known as a "restrictive filling pattern", the E/A ratio is > 2.0, the deceleration time is < 160 ms, and the e/e' ratio is elevated.

Grade IV Diastolic dysfunction: This indicates a poor prognosis and very elevated left atrial pressures. The E/A ratio is > 2.0, the deceleration time is low and the e/e' ratio is elevated. This is rarely seen in cirrhosis.

Albumin related immunological assessment:

Considering immunomodulation as an important mechanism of action of albumin. Additional experiments would be done at baseline, 3 and 6 months to assess the albumin isoforms (HMA, HNA1, HNA2, IMA) , levels of pro-inflammatory and anti-inflammatory cytokines (multiplex luminex based cytokine array) , inflammatory mediators (C-Reactive Protein, endotoxin assay, compliment proteins; DAMPS ); Frequency and functional profile of innate immune cells (monocytes, neutrophills)

Albumin isoforms analysis:

Chemicals Change in albumin isoform will be done by quantification of different albumin modification(HMA, HNA1, HNA2, IMA) on an electron spray ionization orbitrap HRMS system "(Q Exative plus) mass spectrometer coupled to UHPLC from Thermoscientific USA.Briefly the isolated plasma of patients blood at given time point (day 0 and three month) will be diluted with distilled water at a 1:4,000 ratio, and then 8 uL of this diluted plasma will be injected into the high performance liquid chromatography-electron spray ionization MS system. High-performance liquid chromatography separation will be performed on a reverse-phase C8 column (Agilent ZORBAX RRHD 300SB-C8, 2.1 mm id 3 50 mm, 1.8 lm threaded column with a pore size of 300 Å) at a flow rate of 0.2 mL/minute using an H2O-acetonitrile (with 0.1% formic acid) solvent system under a gradient of 90% H2O to 90% acetonitrile over a period of 25 minutes with acquisition starting at 3 minutes. Under auto-MS conditions, mass spectral analysis will be performed. A similar analysis will also be performed with exogenous albumin solution. The obtained compound electron spray ionization MS spectra will be analyzed using the software Protein Deconvolution soft warre (thermoscientific germany). Here, after minimizing the base peak chromatogram from the total ion chromatogram, albumin mass chromatograms will be obtained and analyzed. The obtained albumin spectra will then be deconvoluted within mass range from 66,000-67,000 Da (as the molecular weight [MW] of various albumin isoforms fall within this range. Finally, from the intensity of the peaks, the abundance of albumin isoforms will be measured and the relative abundance of the various HSA isoforms will be reported as described in Das et.al 2017. This will be performed at baseline and 3 months. ( Mass spectrometry (MS)-grade water, acetonitrile, and formic acid will be purchased from Sigma-Aldrich (St. Louis, MO). Purified HSA was purchased from Baxter (Gurgaon, India). All reagents will be of analytical grade.

Cytokine array A panel of 45 cytokines, chemokines, and growth factors will be analyzed in blood plasma of patients group at baseline and 3 months using a Bio-Plex multiplex cytokine bead assay system (Bio-Rad, CA) as per the manufacturer's protocol. The intra-assay and inter assay coefficient of variation considered for multiplex assays will be < 5%

Innate Immune cells profiling:

Total whole blood will be collected from patients pre and post therapy and evaluated for % frequency of monocytes by staining with fluorochrome labeled anti-CD14 anti CD16 and for neutrophils anti-CD11b anti CD16 anti-CD15, anti-CD66b and will acquired and anlaysed using flow cytometry FACS verse (BD biosciences). For the functional profiling of innate immune cells, the blood will be divided into two parts. The PBMCs will be isolated using ficoll-hypaque (Himedia) and monocytes will be isolated using CD14 isolation kit from miltenyi biotech as per the manufacture protocol. Whereas, other part of the blood will be used to isolate the neutrophils using gran-hypaque (Himedia). The intracellular cytokines such as IFN-y, TNF-a, IL-1b will be analysed after low dose of LPS stimulation. Also, phagocytic burst or ROS generation will be done using manufacturer's described protocol. Again the data will be acquired and anlysed using FACS verse (BD biosciences).

Seahorse metabolic analysis methodology:

Effect on energy metabolism of monocytes (that guide the functional property of immune cells) we be analyzed by measuring the extracellular acidification rate (ECAR) and oxygen consumption rate (OCR) through Seahorse XF24 Extracellular Flux Analyzer instrument in peripheral blood monocytes of patients at baseline and 3 months as a measure of lactate production (a surrogate for the glycolytic rate) and OXPHOS respectively. In brief, monocytes will be isolated from freshly collected blood using CD14 isolation kit from miltenyi biotech as per the manufacture protocol. Isolated monocytes will be seeded in triplicate at a density of 1X105 cells per well. Prior to starting the assay, cells will be incubated in Seahorse Assay Medium supplemented with 10 mM glucose and 1 mM sodium pyruvate and glutamine in 37°C incubator without CO2 for 45 min. Further change in parameters of oxidative phosphorylation will be calculated by a real-time change in OCR in response to treatment with Oligomycin (ATPase inhibitor, 1 μM), FCCP (0.2 μM) and rotenone (0.5 μM).

Study Population: Patients with acute decompensation of cirrhosis

Study Design:

* A prospective observational study
* The study will be conducted on patients admitted to Department of Hepatology from 2021-2022
* Study group will comprise of patients of acute decompensation of cirrhosis

Sample Size calculation: Considering the survival benefit with albumin administration as 60% versus 35% with standard medical treatment, the estimated sample size for one-sample comparison of proportion to hypothesized value

Test Ho: p = 0.3500, where p is the proportion in the population

Assumptions:

alpha = 0.0500 (two-sided) power = 0.9500 alternative p = 0.6000

Further, assuming a 20% drop rate

Estimated required sample size:

n = 55 We estimated a minimum sample size of 55 patients for the study.

Intervention: High dose 25% albumin 1.5 gm/kg/week every week for 12 weeks

Monitoring and Assessment: Follow up: every week for 1 month, 2 months and 3 months

Statistical analysis

* All variables shall be expressed in mean (sd) or median (range)
* Variables will be compared by Mann- Whitney U test
* For Categorical variables we will use Chi-Square or Fisher's test
* Survival analysis will be done using Cox-proportional regression analysis
* Actuarial probability of survival shall be calculated by Kaplan- Meier graph and compared by log- rank test.
* Competing risk survival analysis with competing events as TIPS and liver transplant would be performed

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute decompensation of cirrhosis
* Patients with age from 18-65 years

Exclusion Criteria:

* Recent Gastrointestinal bleeding within 7 days
* Patients with organic nephropathy (as defined by IAC)
* Patients with Cardiovascular disease or chronic obstructive pulmonary disease
* Systemic arterial hypertension (>160/90mmhg)
* Presence of hepatocellular carcinoma (outside Milan criteria) ( or portal vein thrombosis
* Budd-Chiari Syndrome
* Pregnancy
* Patients with serum albumin >3 gm
* Refusal to participate
* Known or suspected hypersensitivity to albumin
* Prior TIPS
* Post liver or kidney transplantation
* Patients enrolled in other clinical trials
* Extrahepatic malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute decompensation of cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall mortality. | 3 months

SECONDARY OUTCOMES:
Incidence of liver-related complications. | 1 month
Incidence of liver-related complications. | 3 months
Survival free of liver transplant and TIPS in both groups. | 1 month
Survival free of liver transplant and TIPS in both groups. | 3 months
Delta change in the mean arterial pressure in mm of Hg before and after albumin. | 1 month
  systemic hemodynamics as assessed by the mean arterial pressure in mm of Hg and cardiac function measured by cardiac index from the 2D-Echocardiography in ml/min/m2.
Delta change in the mean arterial pressure in mm of Hg before and after albumin. | 3 months
Delta change coagulation indices measured by the rotational thromboelastometry before and after albumin at 1-month. | 1 month
Delta change coagulation indices measured by the rotational thromboelastometry before and after albumin at 3 months. | 3 months
Delta change in CRP. | 1 months
Delta change in CRP. | 3 months
Delta change in IL-6. | 1 months
Delta change in IL-6. | 3 months
Proportion of patients with reduction in the MELD score by at least 5 points at 1 month. | 1 month
Proportion of patients with reduction in the SOFA score by 2 points at 1 month. | 1 month
Proportion of patients with reduction in the AARC grade by 1 at 1 month. | 1 month
Proportion of patients with reduction in the MELD score by at least 5 points at 3 months. | 3 months
Proportion of patients with reduction in SOFA score by 2 points at 3 months. | 3 months
Proportion of patients with reduction in AARC grade by 1 at 3 months. | 3 months
The cumulative incidence of infections at 1 month. | 1 months
The cumulative incidence of infections at 3 month. | 3 months
Proportion of patients achieving recompensation. | 1 month
Proportion of patients achieving recompensation. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided